CLINICAL TRIAL: NCT02595385
Title: Blood Conservation in Adult Cardiac Surgery, What is the Way Forward in Today's Practice?
Acronym: CONSERVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Alison Murphy, Research Administrator, Belfast Health and Social Care Trust
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 134964
Record Dates: First submitted 2015-10-16; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Adult Cardiac Surgery; Blood Transfusion
MeSH Terms: interventions — Operative Blood Salvage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- RAP (Active Comparator): Retrograde Autologous Prime of the bypass circuit. To remove 500-900ML of fluid.
  Interventions: Procedure: Retrograde Autologous Prime
- CS (Active Comparator): Reinfusion of shed blood during the operation
  Interventions: Device: Cell Salvage
- RAP and CS (Active Comparator): RAP and CS used in combination
  Interventions: Device: Cell Salvage; Procedure: Retrograde Autologous Prime
- Control (No Intervention): No intervention

INTERVENTIONS:
Device: Cell Salvage — Reinfusion of shed blood during the operation
  Arms: CS; RAP and CS
Procedure: Retrograde Autologous Prime — Removal of fluid from the bypass circuit
  Arms: RAP; RAP and CS

SUMMARY:
The aim of this study is to compare retrograde autologous priming (RAP) of the bypass circuit to cell salvage (CS) as part of blood conservation strategies in adult cardiac surgery. It hypothesizes that RAP is at least as effective as cell salvage in terms of blood conservation but at the same time more cost effective.

DETAILED DESCRIPTION:
Cardiac surgery is a major blood consumer. Current evidence shows there is no benefit from transfusion for haematocrits as low as 21% and the risk of death within 30 days of surgery is almost 6 times higher for patients who receive blood. In addition, transfused patients are more likely to experience increased infections and ischaemic complications like myocardial infarction, stroke and renal compromise. While it is agreed to avoid blood transfusion when feasible, there is no current consensus on the best strategy to maintain an acceptable haemocrit and minimise the need for allogenic blood transfusion. Two of the many strategies that have been employed are Retrograde Autologous Prime (RAP) of the bypass circuit and cell salvage (CS) with reinfusion of shed blood.

This study is a prospective, randomised controlled trial with 240 patients undergoing a single procedure adult cardiac surgery that will be randomised to either full crystalloid prime volume or RAP, with or without cell salvage. There will be four study arms;

1. RAP alone
2. Cell Salvage alone
3. RAP plus cell salvage
4. Control group

Results will follow analyse of the data using a logistic regression using a design matric with blood transfused as a key explanatory variable with scope to add in patient covariables. It is expected that date will be analysed after 100 patients and if significance is achieved then the study can be terminated.

The study will aim to identify those patients that receive a blood transfusion intra or post-operatively. Symptomatology from anaemia is subjective and hard to measure. The studies linking transfusion to cardiac surgery outcomes are retrospective; despite careful risk adjustment, it is possible that these associations reflect a tendency amongst clinicians to transfuse the most critically ill patients or miss another important confounder.

In 2001, Spiess referred to current transfusion practice as a 'silent epidemic'. His description is still accurate. In 2006, almost half of all patients undergoing coronary artery bypass grafting in the united states received blood transfusion and the probability of receiving blood is greater when procedures are more complex. Although the infectious risk of blood transfusion have been successfully minimised the weight of evidence increasingly suggests that transfusing less in stable patients could prevent a significant amount of morbidity and mortality. This study will help guide management in those in whom transfusion is avoidable.

ELIGIBILITY:
Inclusion Criteria:

* Less than 80 years of age
* Undergoing single procedure surgery
* Be on single anti-platelet therapy
* To have stopped warfarin pre-operatively with a INR of <1.5
* Have stable coronary disease
* Have good Left Ventricular function

Exclusion Criteria:

* Redo procedures
* Emergency Surgery
* Be on dual antiplatelet therapy
* Have pre-operative kidney dysfunction with eGFR <60ml/min
* Have post-operative drainage >200ml per hour or require re-exploration for bleeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Number of units of packed red blood cells transfused | through study completion, an average of 2 weeks

SECONDARY OUTCOMES:
Adverse reaction to RAP measured by systolic BP <90mmHg during initiation of bypass. | intra-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Reuben Jeganathan, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Department of Medicine, Belfast, United Kingdom